CLINICAL TRIAL: NCT07102901
Title: A Multicenter, Open-Label Phase II Clinical Study Evaluating the Safety, Tolerability and Efficacy of SHR2554 Tablets in Combination With Other Antitumor Therapies in Patients With Locally Advanced Unresectable or Metastatic Gastric or Gastro-oesophageal Junction Adenocarcinoma
Brief Title: Safety and Efficacy of SHR2554 Combined With Other Antitumor Therapies in Gastric or Gastro-oesophageal Junction Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR2554-203-GC
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Advanced Gastric Cancer; Metastatic Gastric Cancer; Gastroesophageal Junction Adenocarcinoma
MeSH Terms: conditions — Stomach Neoplasms | interventions — SHR-1701

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment group A (Experimental)
  Interventions: Drug: SHR2554 Tablets; Drug: SHR-A1811 Injection
- Treatment group B (Experimental)
  Interventions: Drug: SHR2554 Tablets; Drug: SHR-A1904 Injection
- Treatment group C (Experimental)
  Interventions: Drug: SHR2554 Tablets; Drug: SHR-1701 Injection
- Treatment group D (Experimental)
  Interventions: Drug: SHR2554 Tablets

INTERVENTIONS:
Drug: SHR2554 Tablets — Oral SHR2554 tablets.
Drug: SHR-A1811 Injection — SHR-A1811 for injection.
  Arms: Treatment group A
Drug: SHR-A1904 Injection — SHR-A1904 for injection.
  Arms: Treatment group B
Drug: SHR-1701 Injection — SHR-1701 injection
  Arms: Treatment group C

SUMMARY:
This is a multicenter, phase 2, open label study to evaluate safety, tolerability and efficacy of SHR2554 combined with other anti-tumor treatments in patients with advanced or metastatic gastric or gastroesophageal junction adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years or the minimum legal adult age (whichever is greater) at the time the ICF is signed.
2. Has at least 1 measurable lesion based on investigator imaging assessment (computed tomography or magnetic resonance imaging) using RECIST v1.1 at screening.
3. Is willing to provide an adequate tumor sample.
4. Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1 at Screening.

Exclusion Criteria:

1. Presence of dysphagia or other factors impairing oral administration of SHR2554.
2. Has previously been treated with any enhancer of zeste homolog inhibitors.
3. Uncontrolled or significant cardiovascular disease.
4. Has spinal cord compression or clinically active central nervous system metastases, defined as untreated and symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms.
5. Has active autoimmune diseases requiring systemic corticosteroids/immunosuppressants.
6. History of known hypersensitivity to SHR2554 or excipients.
7. Evidence of ongoing uncontrolled systemic bacterial, fungal, or viral infection requiring treatment with intravenous (IV) antibiotics, antivirals, or antifungals.
8. Diagnosis of other malignancies within 5 years prior to the first dose of investigational product.
9. Has history of interstitial lung disease (ILD), non-infectious pneumonitis requiring systemic glucocorticoids, current suspected/confirmed ILD, or clinically significant pulmonary disease history.
10. Psychological, social, familial, or geographical factors that would prevent regular follow-up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs). | Up to approximately 2 years.
  Incidence and severity of adverse events (AEs) graded by Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Incidence and severity of serious adverse events (SAEs). | Up to approximately 2 years.
  Incidence and severity of serious adverse events (SAEs) graded by Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Incidence of Dose Limited Toxicity (DLT). | Up to Day 21.
Objective response rate (ORR) by the investigator assessment. | Up to approximately 1 year.
  Defined as percentage of participants who achieved a best overall response of complete response (CR) or partial response (PR) assessed by the investigator.

SECONDARY OUTCOMES:
Duration of objective tumor response (DoR). | Approximately 24 months.
Disease control rate (DCR). | Approximately 24 months.
Progression-free survival (PFS). | Approximately 24 months.
Overall survival (OS) assessed by the investigator. | Approximately 24 months.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan

IPD SHARING:
Plan to Share IPD: Undecided